CLINICAL TRIAL: NCT01312077
Title: Postoperative Analgesia in Total Hip Replacement: a Comparison of the Analgesic Efficacy of Periarticular Infiltration of Local Anaesthetic With Intrathecal Morphine.
Brief Title: The Analgesic Efficacy of Periarticular Infiltration of Local Anaesthetic for Total Hip Replacement
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cork University Hospital (Other)
Responsible Party: Denise McCarthy, Anaesthesia Specialist Registrar, Cork University Hospital, Cork, Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THR-SMOH
Record Dates: First submitted 2011-03-09; First posted 2011-03-10 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Total Hip Arthroplasty
Keywords: total hip arthroplasty; total hip replacement; local infiltration analgesia; wound infusion; patients undergoing total hip replacement (total hip arthroplasty)
MeSH Terms: interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levobupivacaine infiltration (Experimental): Patients will receive spinal anaesthesia with intrathecal bupivacaine, and will receive peri- and intraarticular surgical site infiltration during surgery and before wound closure with a solution of levobupivacaine 0.5% 2mg/kg body weight with epinephrine made up to a volume of 1.5ml/kg with saline. A catheter will be placed by the surgeon before closure and this will be left in situ in the wound. The catheter will be sited under the fascia lata exiting antero-superior to the incision. A bacterial filter will be attached and it will be connected to an elastomeric pump which will deliver a continuous infusion of levobupivacaine 0.25% at 4ml/hr commencing 6 hours postoperatively and continuing for 24 hours.
  Interventions: Drug: Levobupivacaine
- Control (Other): Patients will receive spinal anaesthesia with intrathecal bupivacaine 0.5% (17.5 mg if greater than 70 kg and 15 mg if less than 70 kg) and preservative-free morphine (0.2 mg).
  Interventions: Drug: Intrathecal morphine

INTERVENTIONS:
Drug: Levobupivacaine — peri- and intraarticular surgical site infiltration before wound closure with a solution of levobupivacaine 0.5% 2mg/kg body weight with epinephrine made up to a volume of 1.5ml/kg with saline. A catheter will be placed by the surgeon before closure under the sterile surgical conditions and this will be left in situ in the wound. An elastomeric pump will deliver a continuous infusion of levobupivacaine 0.25% at 4ml/hr commencing 6 hours postoperatively and continuing for 24 hours.
  Arms: Levobupivacaine infiltration
Drug: Intrathecal morphine — intrathecal morphine bolus 200 micrograms
  Arms: Control

SUMMARY:
Total hip replacement is a major surgical procedure usually associated with significant pain in the early postoperative period. In our hospital, total hip replacement is routinely performed under spinal anaesthesia with intrathecal bupivacaine local anaesthetic plus opioid in the form of preservative free morphine. The use of 'local infiltration analgesia' as an alternative postoperative analgesic technique has been investigated.In this technique the surgeon infiltrates the surgical site with a long-acting local anaesthetic and places a catheter under direct vision which remains in situ and is used to administer local anaesthetic in the postoperative period until such time as it is removed (when no longer deemed necessary for pain relief or at a pre-set time in the postoperative period e.g. 48 hours). We hypothesize that infiltration of the surgical site with peri- and intraarticular levobupivacaine local anaesthetic would be an efficacious pain management technique and would not be inferior to intrathecal morphine for postoperative pain management.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for unilateral total hip replacement
* Consent to spinal anaesthesia
* ASA Grade I to III

Exclusion Criteria:

* Patient refusal
* Mini-Mental Score < 25
* Allergy to bupivacaine, morphine, paracetamol, diclofenac
* Skin lesions/infection at site of injection
* Uncorrected renal dysfunction
* Coagulation disorders
* chronic pain condition other than hip pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Quality of analgesia at 24 hours postoperatively as assessed by visual analogue score (VAS) for pain at rest and on movement. | 24 hours postoperatively

SECONDARY OUTCOMES:
Opioid consumption in the first 48 hours postoperatively. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Denise M McCarthy, MB FCARCSI, Principal Investigator — Cork University Hospital
Locations (1):
- St Mary's Orthopaedic Hospital, Cork, Ireland